CLINICAL TRIAL: NCT04559022
Title: Pilot Study Investigating the Efficacy of Fat Grafting as a Treatment for Male and Female Facial Acne Scarring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey M. Kenkel, Chairman, Department of Plastic Surgery, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 2020-0310
Record Dates: First submitted 2020-09-01; First posted 2020-09-22 (Actual); Results first posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-08

CONDITIONS: Acne Scars - Mixed Atrophic and Hypertrophic; Acne
MeSH Terms: conditions — Hypertrophy; Acne Vulgaris

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fat Grafting for Acne Scar Treatment (Other): This single-center, clinical trial will assess the efficacy and tolerability of the autologous fat grafting when used on men and women with acne scars on the face.
  Interventions: Procedure: Fat Grafting

INTERVENTIONS:
Procedure: Fat Grafting — This single-center, clinical trial will assess the efficacy and tolerability of the autologous fat grafting when used on men and women with acne scars on the face.

SUMMARY:
This single-center, clinical trial consists of a one autologous fat grafting treatment followed by 3-month and 6-month post-treatment visits in order to assess the efficacy of fat grafting when used by men and women with facial acne scars.

DETAILED DESCRIPTION:
This investigation, pilot study will evaluate the safety and efficacy of autologous fat grafting for the treatment of acne scarring. Overall assessment of clinical outcome and safety will be based clinic visits and evaluation of pre- and post- procedural photos. In conjunction with standard and close-up photography, we will also be using 3D imaging, cross-polarized imaging, UV imaging, high-resolution ultrasonography, optical coherence tomography, transepidermal water loss measurements, and/or BTC 2000 measurements. Additionally, we will be utilizing 0.33 mm skin biopsies to assess histological and genetic changes that occur below the skin surface as a result of this treatment. The subject's assessment of satisfaction will be characterized using a non-parametric assessment scale at each follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18 to 50 years of age having general good health.
2. Individuals deemed by the Investigator to have a significant amount acne scarring on the face and that desire correction of this condition.
3. Individuals willing to withhold aesthetic therapies to the areas of the hand being treated or judged to potentially impact results by the Investigator (e.g. soft tissue fillers and/or any resurfacing procedures, botulinum toxin, injectable fillers, microdermabrasion, IPL (intense pulsed light), peels, laser treatments, and tightening treatments, etc.) for the duration of the study. Waxing and threading is allowed but no laser treatments outside of the study.
4. Individuals that are willing to provide written informed consent and are able to read, speak, write, and understand English.
5. Individuals willing to sign a photography release.
6. Willingness to cooperate and participate by following study requirements for the duration of the study and to report any changes in health status or medications, adverse event symptoms, or reactions immediately.

Exclusion Criteria:

1. Individuals diagnosed with known allergies to general skin care products.
2. Individuals who have presence of an active systemic or local skin disease that may affect wound healing.
3. Individuals with sensitivity to topical lidocaine.
4. Individuals who have physical or psychological conditions unacceptable to the Investigator.
5. Individuals who have a recent history of significant trauma to the areas to be treated (< 6 months).
6. Individuals who have severe or cystic active and clinically significant acne on the area(s) to be treated. Clinically significant acne is defined as a subject whom has > 5 active inflammatory acne lesions (including acne conglobate, nodules, or cysts) in either the right or left treatment area.
7. Individuals who have a recent or current history of inflammatory skin disease, infection, unhealed wound or clinically significant acne in the proposed treatment areas.
8. Individuals who have a history of systemic granulomatous diseases, active or inactive, (e.g. Sarcoid, Wegeners, TB, etc.) or connective tissue diseases (e.g. lupus, dermatomyositis, etc.).
9. Individuals who currently have or have a history of hypertrophic scars, or keloid scars.
10. Individuals who currently have cancerous or pre-cancerous lesions in the areas to be treated and/or with a history of skin cancer.
11. Individuals who have the inability to understand instructions or to give informed consent.
12. Individuals who have had microdermabrasion or glycolic acid treatment to the treatment area(s) within one month prior to study participation or who will have this treatment during the study.
13. Individuals who have a history of chronic drug or alcohol abuse.
14. Individuals undergoing concurrent therapy that, in the Investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study device.
15. Individuals who, in the Investigator's opinion, have a history of poor cooperation, noncompliance with medical treatment, or unreliability.
16. Individuals who have a history of the following cosmetic treatments in the area(s) to be treated:

    * Skin tightening procedure within the past year;
    * Injectable filler of any type within the past:

      * 12 months for Hyaluronic acid fillers (e.g. Restylane)
      * 12 months for Ca Hydroxyapatite fillers (e.g. Radiesse)
      * 24 months for Poly-L-Lactic acid fillers (e.g. Sculptra)
      * Ever for permanent fillers (e.g. Silicone, ArteFill)
    * Neurotoxins within the past three months;
    * Ablative resurfacing laser treatment;
    * Non-ablative, rejuvenative laser or light treatment within the past six months;
    * Surgical dermabrasion;
    * Had a chemical peel or dermabrasion, of the dorsum of the hand within four weeks
17. Individuals with a history of using the following prescription medications:

    * Accutane or other systemic retinoids within the past six months;
    * Topical Retinoids within the past two weeks;
    * Prescription strength skin lightening devices (e.g. hydroquinone, tretinoin, AHA, BHA and polyhydroxy acids, 4-hydroxyanisole alone or in combination with tretinoin, etc.) within four months;
    * Any anti-wrinkle, skin lightening devices, or any other device or topical or systemic medication known to affect skin aging or dyshcromia (devices containing alpha/beta/poly-hydroxy acids, vitamin C, soy, Q-10, hydroquinone; systemic or licorice extract (topically), Tego® Cosmo C250, gigawhite, lemon juice extract (topically), emblica extract, etc.) within two weeks;
    * Antiplatelet agents/Anticoagulants (Coumadin, Heparin, Plavix, chronic NSAID use); and/or
    * Psychiatric drugs that in the Investigator's opinion would impair the subject from understanding the protocol requirements or understanding and signing the informed consent.
18. Individuals who are nursing, pregnant, or planning to become pregnant during the study according to subject self-report.
19. Individuals having a health condition and/or pre-existing or dormant dermatologic disease on the body (e.g., psoriasis, rosacea, eczema, seborrheic dermatitis, vitiligo, hyper or hypo-skin pigmentation conditions such as post inflammatory hyperpigmentation) that the Investigator or designee deems inappropriate for participation or could interfere with the outcome of the study.
20. Individuals with a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications (e.g., azathioprine, belimumab, cyclophosphamide, Enbrel, Imuran, Humira, mycophenolate mofetil, methotrexate, prednisone, Remicade, Stelara.) and/or radiation as determined by study documentation.
21. Individuals with an uncontrolled disease such as asthma, diabetes, hyperthyroidism, medically significant hypertension or hypothyroidism. Individuals having multiple health conditions may be excluded from participation even if the conditions are controlled by diet, medication, etc.
22. Individuals with any planned surgeries, overnight hospitalization, and/or invasive medical procedures during the course of the study.
23. Individuals who have observable suntan, nevi, excessive hair, etc. or other dermal conditions on the back of the hand that might influence the test results in the opinion of the Investigator or designee.
24. Individuals who have any condition, which in the opinion of the Investigator makes the patient unable to complete the study per protocol (e.g. patients not likely to avoid other cosmetic treatments to the treatment area; patients not likely to stay in the study for its duration because of other commitments, concomitant conditions, or past history; patients anticipated to be unreliable, or patients who have a concomitant condition that may develop symptoms that might confuse or confound study treatments or assessments).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Kenkel, MD, Principal Investigator — UT Southwestern
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fat Grafting for Acne Scar Treatment
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fat Grafting for Acne Scar Treatment
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 1
  Unknown or Not Reported | 0
Fitzpatrick Skin Score [Count of Participants; unit: Participants] — The Fitzpatrick scale is a numerical classification schema for human skin color to estimate response of skin to UV light.
  Fitzpatrick type & Characteristics
  1. always burns, never tans (palest; freckles)
  2. usually burns, tans minimally (light colored but darker than pale)
  3. sometimes mild burn, tans uniformly (golden honey or olive)
  4. burns minimally, always tans well (moderate brown)
  5. very rarely burns, tans very easily (dark brown)
  6. never burns (deeply pigmented dark brown to darkest brown)
  Participants
    Type 1 | 0
    Type 2 | 6
    Type 3 | 1
    Type 4 | 3
    Type 5 | 0
    Type 6 | 0

OUTCOME MEASURES:

1. Primary Outcome: Subject Acne Severity Scale
Description: The Goodman and Baron Qualitative Acne Scale will be used to assess acne scars.
  Grade 1- Macular Disease: Erythematous, hyper- or hypopigmented flat marks Grade 2- Mild Disease: Mild rolling, small soft papular Grade 3- Moderate Disease: More significant rolling, shallow "box car", mild to moderate hypertrophic or papular scars Garde 4- Severe disease: Punched out atrophic, "ice pick", bridges and tunnels, gross atrophy, dystrophic, scars significant hypertrophy or keloid
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Fat Grafting for Acne Scar Treatment
Number analyzed (Participants) | 10
Participants
  Grade 1: Macular | 0
  Grade 2: Mild | 1
  Grade 3: Moderate | 2
  Grade 4: Severe | 7

2. Primary Outcome: Facial Photograph Assessments- Global Aesthetic Improvement Scale
Description: Subjects and Clinicians will evaluate efficacy of treatment at follow up visits. The photographs from follow up visits will be compared to their baseline photographs.
  Acne scars on patients will be assessed using the Global Aesthetic Improvement Scale by subject and clinician.
  CGAIS Rating
  1. Very much improved: Optimal cosmetic result.
  2. Much improved: Marked improvement in appearance from the initial condition, but not completely optimal.
  3. Improved: Obvious improvement in appearance from initial condition.
  4. No Change: The appearance is essentially the same as the original condition.
  5. Worse: The appearance is worse than the original condition.
Time Frame: Month 3 and Month 6
Measure: Median (Standard Error); unit: units on a scale
Groups:
- In Person Subject Assessment: S-GAIS was completed by subject at follow up visits (Month 3 and Month 6 post treatment)
- Clinician Assessment: The Clinician GAIS was completed after study completion.
Arm/Group | In Person Subject Assessment | Clinician Assessment
Number analyzed (Participants) | 10 | 10
units on a scale
  Month 3 | 2.7 (.36) | 3 (.37)
  Month 6 | 2.8 (.26) | 3.2 (.25)

3. Primary Outcome: Topographical Analysis of Texture
Description: MiraVex will be used to assess changes in texture (roughness) of the subjects facial acne scars.
Time Frame: Baseline and 6 Months
Measure: Mean (Standard Error); unit: mm
Groups:
- Baseline; Month 6: This single-center, clinical trial will assess the efficacy and tolerability of the autologous fat grafting when used on men and women with acne scars on the face.
  Fat Grafting: This single-center, clinical trial will assess the efficacy and tolerability of the autologous fat grafting when used on men and women with acne scars on the face.
Arm/Group | Baseline | Month 6
Number analyzed (Participants) | 10 | 10
mm
  Maximum Depth of Depressions (mm) | 0.1495 (0.019) | 0.0536 (0.017)
  Roughness (Ra) | 17.55 (1.5) | 16.58 (1.6)

4. Primary Outcome: Histological Analysis
Description: Relative changes in protein abundance in biopsies taken at post treatment compare to control or entreated group will be quantified using an image processing software based on fluorescence signal intensity. The change from baseline was calculated at each time frame.
Time Frame: Baseline, 3 Months and 6 Months
Measure: Mean (Standard Error); unit: percentage change from baseline
Groups:
- Papillary Dermis- Type I Collagen; Papillary Dermis- Type III Collagen; Reticular Dermis- Type I Collagen; Reticular Dermis- Type III Collagen: Microbiopsies were collected at baseline and follow up visits. Analysis was used to correlate changes seen with noninvasive skin measurements and clinical assessment with histological changes in ultrastructure.
Arm/Group | Papillary Dermis- Type I Collagen | Papillary Dermis- Type III Collagen | Reticular Dermis- Type I Collagen | Reticular Dermis- Type III Collagen
Number analyzed (Participants) | 10 | 10 | 10 | 10
percentage change from baseline
  Baseline | 1.00 (0.09) | 1.00 (.25) | 1.0 (.18) | 1.0 (.26)
  Month 3 | 1.07 (0.13) | 0.87 (0.24) | 0.76 (0.10) | 0.74 (0.08)
  Month 6 | 0.85 (0.05) | 0.76 (0.15) | 0.85 (0.06) | 0.62 (0.13)

5. Primary Outcome: Gene Expression
Description: Biopsies of the treated are will be taken prior to treatment and post treatment for gene expression analysis. This analysis will identify gene expression related to collagen formation and increased cell turnover.
Time Frame: Baseline, 3 Months and 6 Months
Measure: Mean (Standard Error); unit: percentage change from baseline
Groups:
- Type 1 Collagen; Type III Collagen; Elastin; Lysl Oxidase; Matrix Metalloproteinase-2; Tissue Growth Factor B1; Tissue Growth Factor B3: Relative changes in protein abundance in biopsies taken at post treatment compare to control or entreated group will be quantified using an image processing software based on fluorescence signal intensity. The change from baseline was calculated at each time frame.
Arm/Group | Type 1 Collagen | Type III Collagen | Elastin | Lysl Oxidase | Matrix Metalloproteinase-2 | Tissue Growth Factor B1 | Tissue Growth Factor B3
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10
percentage change from baseline
  Baseline | 1.13 (0.20) | 1.21 (0.34) | 1.31 (0.49) | 1.46 (0.58) | 1.17 (0.24) | 1.19 (0.32) | 1.37 (0.55)
  Month 3 | 1.48 (0.83) | 1.68 (1.00) | 0.45 (0.19) | 0.69 (0.32) | 0.66 (0.28) | 0.65 (0.07) | 0.40 (0.01)
  Month 6 | 0.58 (0.13) | 0.58 (0.12) | 0.59 (0.27) | 0.53 (0.12) | 0.43 (0.12) | 0.61 (0.12) | 0.56 (0.14)

6. Secondary Outcome: Noninvasive Skin Assessments- TEWL
Description: Transepidermal Water Loss (TEWL) was measured at baseline and 6 months after treatment.
Time Frame: Month 3 and Month 6
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Groups:
- 3-Month Follow Up; 6-Month Follow Up: This single-center, clinical trial will assess the efficacy and tolerability of the autologous fat grafting when used on men and women with acne scars on the face.
  Fat Grafting: This single-center, clinical trial will assess the efficacy and tolerability of the autologous fat grafting when used on men and women with acne scars on the face.
Arm/Group | 3-Month Follow Up | 6-Month Follow Up
Number analyzed (Participants) | 10 | 10
percentage change from baseline | 8.74 (3.41) | 35.37 (11.18)

7. Secondary Outcome: Noninvasive Skin Assessments- High-resolution Ultrasonography
Description: Ultrasonography was used to measure epidermal/dermal thickness/density 3 and 6 months after treatment.
  Percent change from baseline results are reflected.
Time Frame: Month 3 and Month 6
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | 3-Month Follow Up | 6-Month Follow Up
Number analyzed (Participants) | 10 | 10
percentage change from baseline
  Epidermal Thickness | -4.28 (12.37) | -0.63 (10.98)
  Epidermal Density | 21.34 (22.05) | -2.9 (11.96)
  Dermal Thickness | -26.4 (212.46) | -19.4 (330.59)
  Dermal Density | 53.5 (11.248) | -12.9 (5.41)

8. Secondary Outcome: Noninvasive Skin Assessments- Skin Deformation
Description: biomechanical analysis of skin deformation was used to measure skin laxity, skin elasticity, viscoelastic deformation, ultimate deformation, stiffness and energy absorption at 3 and 6 months after treatment.
  Percent change from baseline results are reflected.
Time Frame: Month 3 and Month 6
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | 3-Month Follow Up | 6-Month Follow Up
Number analyzed (Participants) | 10 | 10
percentage change from baseline
  Skin Laxity | -5.88 (0.33) | -5.16 (0.36)
  Skin Elasticity | 7.36 (0.18) | -5.62 (0.34)
  Viscoelastic Deformation | 3.57 (0.03) | 2.38 (0.34)
  Ultimate Deformation | -6.90 (0.25) | -11.61 (0.35)
  Stiffness | -1.53 (46.22) | 4.05 (49.68)
  Energy Absorption | -2.35 (11.30) | -6.07 (0.820)

9. Primary Outcome: Topographical Analysis of Depressions
Description: MiraVex will be used to assess changes in depressions of the subjects facial acne scars.
Time Frame: Baseline and 6 Months
Measure: Mean (Standard Error); unit: mm^3
Arm/Group | Baseline | Month 6
Number analyzed (Participants) | 10 | 10
mm^3 | 11.45 (2.36) | 10.64 (2.4)

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Fat Grafting for Acne Scar Treatment
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fat Grafting for Acne Scar Treatment (N=10)
Covid (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT04559022/Prot_SAP_000.pdf